CLINICAL TRIAL: NCT01779141
Title: A Multi-center Observational Study During Pregnancy for Women With T1DM Treated With the Paradigm Insulin Pumps Donated by the 'Wielka Orkiestra Świątecznej Pomocy' Foundation in Poland
Brief Title: Orchestra Pregnancy Observational Study in Poland
Status: Completed | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Collaborators: Medtronic Poland Spółka z ograniczoną odpowiedzialnością (Industry)
Responsible Party: Sponsor
Other Study IDs: PL01
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes Mellitus; Pregnancy
Keywords: Type 1 Diabetes Mellitus - T1DM; Pregnancy; Insulin Pump; Glucose Sensor; Continuous Subcutaneous Insulin Infusion - CSII; Sensor Augmented Pump - SAP; Continuous Glucose Monitoring - CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Biospecimen Retention: None Retained — Whole blood, serum, urine samples as required in routine practice before, during and after pregnancy in women with Type 1 Diabetes Mellitus
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CSII: Patients using CSII with or without CGM.

SUMMARY:
The aim of this project is to document the use of insulin pump therapy (CSII), including sensor augmented pump therapy (SAP), before, during and after pregnancy in women with type 1 Diabetes Mellitus benefiting from the Orchestra donation of Paradigm REAL-Time and Paradigm Veo pumps in Poland.

DETAILED DESCRIPTION:
The project is designed as a multi-center prospective observational Post-Market-Release study to be conducted in up to 30 centers in Poland.

Total duration of the study per patient will be up to 22 months (up to 12 months pre-conception phase, pregnancy, and 6 weeks after delivery). The optimal study start is the beginning of pre-conception phase, however, pregnant women up to the 16th week of pregnancy can participate in the study too. The study end is 6 weeks after delivery. If conception does not occur within 12-months, the patient's study participation is terminated, and the insulin pump might be taken away from the patient. The following therapy is decided by the investigator. If the pump is not taken away after the 12-month of trial period for conception, the patient can continue insulin pump therapy until the pump is needed for another patient.

ELIGIBILITY:
Inclusion Criteria:

1. Female diagnosed with Diabetes Mellitus Type 1
2. Subject indicated by HCP to start insulin pump therapy (CSII) or sensor augmented pump therapy (SAP) due to the desired or established pregnancy
3. HCP has prescribed the use of Orchestra donated device to the subject independently of the study
4. Signed Patient Informed Consent (PIC)
5. Subject is 18 to 45 years old, planning immediate pregnancy (within the next 12 months) or being pregnant within the first trimester until the 16th week of amenorrhea
6. Subject has been on MDI for at least 3 months before starting pump therapy

Exclusion Criteria:

1. Subject was enrolled in the registry earlier, and terminated it (for any reason)
2. Participation in any other interventional clinical trial - currently and/or in the last 3 months before the signature of PIC
3. Subject uses an insulin pump that was not donated by the Orchestra Foundation
4. Pregnant women with longer than 16 weeks of pregnancy/amenorrhea
5. Subjects who need assisted in vitro fertilization
6. Subjects with Diabetes Mellitus Type 2, Gestational Diabetes, MODY or any other type of diabetes than Type 1
7. Subject under the age of 18
8. Subject legally incompetent
9. Subject cannot read or write

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study subject population is women with Type 1 Diabetes Mellitus at the age of 18-45 who
  * plan pregnancy
  * are in the early phase of pregnancy, up to the 16th week
Sampling Method: Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2013-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Sieradzki, Prof, Study Chair — Cracow Medical University
Locations (24):
- Poland (24):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - NZOZ Specjalistyczny Ośrodek Internistyczno-Diabetologiczny, Bialystok
  - Szpital Wojewódzki w Bielsku Białej, Bielsko-Biala
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Szpital Specjalistyczny w Jaśle, Jasło
  - NZOZ WITAMED Outpatient Diabetes Clinic, Kielce
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Łodzi, Lodz
  - Uniwersytet Medyczny w Łodzi, Klinika Diabetologii, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 Uniwersytetu Medycznego w Lublinie, Lublin
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - PSZOZ Wojewódzkie Centrum Medyczne w Opolu, Opole
  - Clinic of Gynecology and Obstetrics of Marcinkowski Medical University, Poznan
  - Zakład Opieki Zdrowotnej Poznań-Jeżyce, Poznan
  - Szpital Wojewódzki nr 2 im. Św. Jadwigi Królowej, Rzeszów
  - Samodzielny Publiczny Wojewódzki Szpital Zespolony w Szczecinie im. Marii Skłodowskiej-Curie, Szczecin
  - Wojewódzki Szpital Zespolony im. L. Rydygiera, Torun
  - Szpital Kliniczny im. ks. Anny Mazowieckiej Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw
  - Mazowiecki Szpital Wojewódzki Sp. z o.o., Warsaw
  - Wojewódzki Zespół Specjalistycznej Opieki Zdrowotnej, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im prof. Stanisława Szyszko, Zabrze
  - Zespół Wojewódzkich Przychodni Specjalistycznych w Katowicach, Zabrze
  - NZOZ MED-ART Poradnie Specjalistyczne Sp. z o.o., Żory

REFERENCES:
- [Derived] Cypryk K, Wender-Ozegowska E, Cyganek K, Sieradzki J, Skoczylas K, Chen X, Cordero TL, Shin J, Cohen O. Insulin pump therapy with and without continuous glucose monitoring in pregnant women with type 1 diabetes: a prospective observational Orchestra Foundation study in Poland. Acta Diabetol. 2023 Apr;60(4):553-561. doi: 10.1007/s00592-022-02020-9. Epub 2023 Jan 19. PMID 36653533

RESULTS

PARTICIPANT FLOW:
Groups:
- CSII: Patients using CSII, with or without CGM
Period: Overall Study
Arm/Group | CSII
Started | 481
Completed | 300
Not Completed | 181

BASELINE CHARACTERISTICS:
Arm/Group | CSII
Number analyzed (Participants) | 481
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 481
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.42 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 481
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 481

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Changes in HbA1C from baseline to after delivery.
Time Frame: from preconception phase to 6 weeks after delivery
Population: Participants who have both baseline HbA1C and after delivery HbA1C available.
Measure: Mean (Standard Deviation); unit: HbA1C percentage
Arm/Group | CSII
Number analyzed (Participants) | 219
HbA1C percentage | -0.8 (1.0)

2. Primary Outcome: Percent of Sensor Glucose Values in 70-140 mg/dL
Description: Percent of sensor glucose values between and including 70 mg/dL to 140 mg/dL
Time Frame: During pregnancy
Population: Subjects with sensor information during pregnancy
Measure: Mean (Standard Deviation); unit: percentage of available sensor values
Arm/Group | CSII
Number analyzed (Participants) | 190
percentage of available sensor values | 67.62 (10.59)

3. Secondary Outcome: Large for Gestational Age (LGA)
Description: Percentage of mothers who delivered LGA babies. The Babies whose weight were greater than 90th percentiles at the gestational age when they were born, were defined as LGA Babies. (reference: Fetal biometry between 20-42 weeks of gestation for Polish population).
Time Frame: after birth
Population: Participants who delivered live babies
Measure: Count of Participants; unit: Participants
Arm/Group | CSII
Number analyzed (Participants) | 320
Participants | 74

4. Secondary Outcome: Unhealthy Babies
Description: The number of participants who delivered babies classified as large for gestational age, with congenital malfunction, or who required mechanical ventilation.
Time Frame: from birth to 6 weeks after delivery
Population: Participants who delivered alive babies
Measure: Count of Participants; unit: Participants
Arm/Group | CSII
Number analyzed (Participants) | 320
Participants | 99

ADVERSE EVENTS:
Time Frame: from preconception phase, throughout pregnancy, during delivery and after delivery during lactation phase (up to 6 weeks), up to 22 months in total per subject
Arm/Group | CSII
All-Cause Mortality (participants affected / at risk) | 1/481
Serious Adverse Events (participants affected / at risk) | 181/481
Other Adverse Events (participants affected / at risk) | 11/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSII (N=481)
Fetal heart rate disorder (Cardiac disorders) | 1 (1)
Truncus arteriosus persistent (Congenital, familial and genetic disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 28 (28)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 5 (5)
Amniotic cavity infection (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Anaemia neonatal (Blood and lymphatic system disorders) | 2 (2)
Apgar score low (Investigations) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 2 (2)
Bradycardia foetal (Cardiac disorders) | 1 (1)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Caesarean section (Surgical and medical procedures) | 11 (11)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 5 (5)
Cervical polyp (Reproductive system and breast disorders) | 1 (1)
Cholestasis of pregnancy (Hepatobiliary disorders) | 2 (2)
Cholestasis of pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Cleft Palate (Congenital, familial and genetic disorders) | 1 (1)
Colloid brain cyst (Nervous system disorders) | 1 (1)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 2 (2)
Congenital infection (Congenital, familial and genetic disorders) | 1 (1)
Congenital pneumonia (Congenital, familial and genetic disorders) | 6 (6)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 (8)
Diabetic eye disease (Eye disorders) | 1 (1)
Diabetic gastropathy (Gastrointestinal disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2)
Diabetic retinopathy (Eye disorders) | 1 (1)
Duodenogastric reflux (Gastrointestinal disorders) | 1 (1)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 1 (1)
Foetal cardiac disorder (Cardiac disorders) | 1 (1)
Foetal disorder (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 17 (18)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Foetal heart rate abnormal (Investigations) | 1 (1)
Foetal heart rate decreased (Investigations) | 4 (6)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 6 (7)
Foetal malformation (Congenital, familial and genetic disorders) | 1 (1)
Foetal monitoring abnormal (Investigations) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 3 (4)
Haemorrhage (Vascular disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 3 (3)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Vascular disorders) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (8)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 1 (1)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Intrauterine infection (Infections and infestations) | 2 (2)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 27 (27)
Ketoacidosis (Metabolism and nutrition disorders) | 2 (2)
Kidney malformation (Congenital, familial and genetic disorders) | 1 (1)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Low birht weight baby (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Maternal condition affecting foetus (Pregnancy, puerperium and perinatal conditions) | 4 (4)
Microtia (Congenital, familial and genetic disorders) | 1 (1)
Neinatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neonatal infection (Infections and infestations) | 3 (3)
Neonatal pneumonia (Infections and infestations) | 5 (5)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oedema (General disorders) | 1 (1)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Ophthalmia neonatorum (Infections and infestations) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 8 (8)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 26 (26)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 6 (6)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal aplasia (Congenital, familial and genetic disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (2)
Reproductive tract and breast procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Tachycardia foetal (Cardiac disorders) | 3 (3)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 17 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ultrasound Doppler abnormal (Investigations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Urinary tract infection neonatal (Infections and infestations) | 1 (1)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Uterine rupture (Injury, poisoning and procedural complications) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 2 (2)
Viral diarrhoea (Infections and infestations) | 1 (1)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSII (N=481)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Caesarean section (Surgical and medical procedures) | 1 (1)
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Congenital pulmonary artery anomaly (Congenital, familial and genetic disorders) | 1 (1)
Ectopic kidney (Congenital, familial and genetic disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Neonatal pneumonia (Infections and infestations) | 1 (1)
Retinopathy haemorrhagic (Eye disorders) | 1 (1)
Umbilical cord vascular disorder (Pregnancy, puerperium and perinatal conditions) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT01779141/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT01779141/SAP_001.pdf